CLINICAL TRIAL: NCT02722161
Title: A Phase I, Open-label, Single-dose Trial to Investigate Metabolism and Pharmacokinetics of [14C]BI 1482694 Administered as Oral Solution in Healthy Male Volunteers
Brief Title: Olmutinib (BI 1482694) ADME Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1370.7; 2016-000190-20 (EudraCT Number: EudraCT)
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Healthy

ARMS (1):
- [14C]BI 1482694 (Experimental)
  Interventions: Drug: [14C]BI 1482694

INTERVENTIONS:
Drug: [14C]BI 1482694

SUMMARY:
To investigate the basic pharmacokinetics of BI 1482694, its metabolites M1 and M2, and [14C]-radioactivity, including mass balance, excretion pathways and metabolism following a single oral dose of [14C]BI 1482694 given to healthy male volunteers

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP [Blood Pressure], PR [Pulse Rate]), 12-lead ECG (Electrocardiogram), and clinical laboratory tests
* Age of 45 to 65 years (incl.)
* BMI (Body Mass Index) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Subjects who are sexually active must use, with their partner, highly effective contraception from the time of administration of trial medication until 4 months after administration of trial medication. Adequate methods are:
* Condoms plus use of hormonal contraception by the female partner that started at least 2 months prior to administration of trial medication (e.g., implants, injectables, combined oral or vaginal contraceptives, intrauterine device) or
* Condoms plus surgical sterilization (vasectomy at least 1 year prior to enrolment) or
* Condoms plus surgically sterilised partner (including hysterectomy) or
* Condoms plus intrauterine device or
* Condoms plus partner of non-childbearing potential (including homosexual men) Subjects are required to use condoms to prevent unintended exposure of the partner to the study drug via seminal fluid. Male and female condoms must not be used together. Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, with their partner, they must comply with the contraceptive requirements detailed above.

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Clinically significant gastrointestinal, hepatic, renal, respiratory (including but not limited to interstitial lung disease), cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/heart rate-corrected QT interval
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
* Smoker (more than 5 cigarettes or 1 cigar or 1 pipe per day)
* Inability to refrain from smoking on specified trial days
* Average intake of more than 24 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/heart rate-corrected QT interval (such as heart rate-corrected QT intervals following the formula of Fridericia that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 10 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
* Irregular defecation pattern (less than a mean of one bowel movement a day)
* Platelet count < 100 * 10^9 cells/L

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of [14C]-radioactivity in urine: fe urine, 0-tz (fraction excreted in urine as percentage of the administered dose over the time interval from 0 to the last quantifiable time point) | up to 1181 hours (7 weeks)
Mass balance recovery of [14C]-radioactivity in faeces: fe faeces, 0-tz (fraction excreted in faeces as percentage of the administered dose over the time interval from 0 to the last quantifiable time point) | up to 1181 hours (7 weeks)

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte) for BI 1482694 in plasma | up to 72 hours
Cmax (maximum measured concentration of the analyte) for [14C]-radioactivity in plasma | up to 336 hours
AUC0-tz (area under the concentration-time curve of the analyte over the time interval from 0 to the last quantifiable time point) for BI 1482694 in plasma | up to 72 hours
AUC0-tz (area under the concentration-time curve of the analyte over the time interval from 0 to the last quantifiable time point) for [14C]-radioactivity in plasma | up to 336 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1370.7.31001 Boehringer Ingelheim Investigational Site, Zuidlaren, Netherlands